CLINICAL TRIAL: NCT00657553
Title: Preemptive Strike With Bortezomib (VELCADE) in Participants With Multiple Myeloma Still Event-free on Total Therapy 2 (UARK 98-026)
Brief Title: Preemptive Strike With Bortezomib in Multiple Myeloma Patients
Acronym: 2007-77
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100241
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bortezomib/Treatment Arm (Active Comparator): Bortezomib Maintenance Year 1 - bortezomib days 1, 4, 8, 11 every 28 days Year 2 - bortezomib days 1, 4, 8, 11 every 2 months Year 3 - bortezomib days 1, 4, 8, 11 every 3 months
  Interventions: Drug: Bortezomib
- Observation Arm (watchful waiting) (No Intervention): monitor myeloma parameters every 3-6 months

INTERVENTIONS:
Drug: Bortezomib — Year 1:1.0 mg/m2. IV. Days 1, 4, 8, 11 every 4 weeks Year 2: 1.0 mg/m2. IV. Days 1, 4, 8, 11 every 8 weeks Year 3: 1.0 mg/m2. IV. Days 1, 4, 8, 11 every 12 weeks
  Other Names: Velcade
  Arms: Bortezomib/Treatment Arm

SUMMARY:
To evaluate whether using the drug bortezomib at the start of remission will prevent relapse for a longer period of time.

DETAILED DESCRIPTION:
Although advances in the treatment of multiple myeloma have led to improved remission rates, the risk for serious relapse is very high. The drug Bortezomib has been highly effective for treatment of the disease in an advanced stage such as post-transplant relapse. Due to the need of maintenance therapies, it is necessary to look to certain drugs that may prolong remission and increase the quality of life. Bortezomib, when taken at the beginning of remission, may prove to be a beneficial maintenance drug for the management of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple myeloma currently or previously enrolled on UARK 98-026 and currently event-free at the time of the evaluation.
* Performance status of 0-2 based of Southwest Oncology Group (SWOG) criteria
* Previously documented platelet count > 75,000/ul within a 35 days prior to enrollment
* Previously documented peripheral absolute neutrophil count >1,000/ul within 35 days prior to enrollment.
* Adequate renal function
* Signed informed consent
* Female subject is post-menopausal or willing to use acceptable birth control
* Male subjects agree to use acceptable method of contraceptive

Exclusion Criteria:

* Hypersensitivity to Bortezomib, boron, or mannitol
* Female subject is pregnant or breastfeeding
* Experienced myocardial infraction within 6 months prior to enrollment
* Received other investigational new drugs within 14 days before enrollment
* Received any anti-myeloma therapy within 14 days
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 3 years of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Myeloma Institute for Research and Therapy, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Bortezomib will be administered as 12 monthly courses of 1.0 mg/m2 on days 1, 4, 8, and 11 and repeated every 28 days, followed by cycles administered every other month in year 2, and then every 3 months in year 3
- Observation Arm: Patients will be observed for progress over the course of three years.
Period: Overall Study
Arm/Group | Treatment Arm | Observation Arm
Started | 5 | 5
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — low accrual, no analysis run | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Observation Arm | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.89) | 64.4 (7) | 63 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Effect of Maintenance Therapy With Bortezomib on the Length of Remission in Participants Currently Receiving Maintenance Therapy as Part of Total Therapy 2
Description: The number of patients on Bortezomib that have maintained event-free survival, compared to the patients on observation was not analyzed due to low attrition rates.
  Event-free survival is a measure of the proportion of people who remain free of a particular complication of disease (called an event) after treatment that is designed to prevent or delay that particular complication.
Time Frame: three years
Arm/Group | Treatment Arm | Observation Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: there were no events reported in the five participants enrolled in the treatment arm or in the five participants enrolled in the observation arm of this study.
Arm/Group | Treatment Arm | Observation Arm
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No